CLINICAL TRIAL: NCT02623296
Title: A Phase I, Drug-drug Interaction Study Between Oral Doses of GLPG1205 and a Cocktail of CYP2C9, CYP2C19 and CYP1A2 Substrates in Healthy Male Subjects
Brief Title: A Drug-drug Interaction Study Between GLPG1205 and a Cocktail of CYP450 Substrates in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1205-CL-103; 2015-002785-23 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG1205 and single CYP450 substrate cocktail dose (Experimental): Daily GLPG1205 administration from Day 1 to Day 12 Single GLPG1205 co-administration on Day 13 with CYP450 substrate cocktail
  Interventions: Drug: GLPG1205; Drug: Cocktail of CYP450 substrates
- Placebo and single CYP450 substrate cocktail dose (Placebo Comparator): Daily Placebo administration from Day 1 to Day 12 Single Placebo co-administration on Day 13 with CYP450 substrate cocktail
  Interventions: Drug: Placebo; Drug: Cocktail of CYP450 substrates

INTERVENTIONS:
Drug: GLPG1205 — Once daily administration of 2 GLPG1205 capsules from Day 1 to Day 13
  Arms: GLPG1205 and single CYP450 substrate cocktail dose
Drug: Placebo — Once daily administration of 2 matching placebo capsules from Day 1 to Day 13
  Arms: Placebo and single CYP450 substrate cocktail dose
Drug: Cocktail of CYP450 substrates — Single administration on Day 13 of cocktail of CYP450 substrates: warfarin tablet, omeprazole capsule and caffeine oral solution

SUMMARY:
This will be a Phase I, randomized, double-blind, placebo-controlled, 2 period cross-over, drug-drug interaction study to evaluate the effect of multiple oral doses of GLPG1205 or placebo (daily from Day 1 to Day 12) on a single dose pharmacokinetic profile of a cocktail of CYP450 substrates administered to healthy male subjects. The cocktail of CYP450 substrates will consist of 10 mg warfarin (CYP2C9 substrate), 20 mg omeprazole (CYP2C19 substrate) and 100 mg caffeine (CYP1A2 substrate).

Fourteen healthy male subjects will receive during two treatment periods from Day 1 to Day 12 a daily dose of GLPG1205 or placebo. On Day 13, a single dose of the cocktail of CYP450 substrates will be co-administered either with GLPG1205 or with placebo. The two treatment periods will be separated by a wash-out period of at least 28 days.

Also, the safety and tolerability of multiple oral doses of GLPG1205 administered with or without a cocktail of CYP450 substrates in healthy male subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Poor or moderate metabolizer for CYP2C9 or CYP2C19 as determined by genotyping
* Having a contraindication as indicated in the respective Summary of Product Characteristics (or Package Leaflets) for warfarin, omeprazole or caffeine
* Intake of nutraceuticals within 3 weeks prior to dosing or within 6 times the elimination half life
* Intake of enzyme inducing or enzyme inhibiting drugs within 3 months prior to dosing
* Intake of vitamin K within 3 weeks prior to dosing
* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The maximum observed concentration (Cmax) of CYP450 substrates in plasma after multiple oral doses of GLPG1205 or placebo | Between Day 13 and 7 days after the last dose
  To characterize the maximum observed concentration (Cmax) of CYP450 substrates in plasma over time after a single dose of a cocktail of CYP450 substrates and multiple doses of GLPG1205 or placebo in healthy male subjects
The time of occurrence of Cmax (tmax) of CYP450 substrates in plasma after multiple oral doses of GLPG1205 or placebo | Between Day 13 and 7 days after the last dose
  To characterize the time of occurrence of Cmax (tmax) of CYP450 substrates in plasma after a single dose of a cocktail of CYP450 substrates and multiple doses of GLPG1205 or placebo in healthy male subjects
The area under the plasma concentration versus time curve (AUC) of CYP450 substrates in plasma after multiple oral doses of GLPG1205 or placebo | Between Day 13 and 7 days after the last dose
  To characterize the area under the plasma concentration versus time curve (AUC) of CYP450 substrates in plasma after a single dose of a cocktail of CYP450 substrates and multiple doses of GLPG1205 or placebo in healthy male subjects
The apparent terminal half-life (t1/2) of CYP450 substrates in plasma after multiple oral doses of GLPG1205 or placebo | Between Day 13 and 7 days after the last dose
  To characterize the apparent terminal half-life (t1/2) of CYP450 substrates in plasma after a single dose of a cocktail of CYP450 substrates and multiple doses of GLPG1205 or placebo in healthy male subjects
The metabolite over parent AUC ratio (R) of CYP450 substrates in plasma after multiple oral doses of GLPG1205 or placebo | Between Day 13 and 7 days after the last dose
  To characterize the metabolite over parent AUC ratio (R) of CYP450 substrates in plasma after a single dose of a cocktail of CYP450 substrates and multiple doses of GLPG1205 or placebo in healthy male subjects

SECONDARY OUTCOMES:
Number of adverse events | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of the number of adverse events reported
Changes in vital signs as measured by heart rate, blood pressure, respiratory rate and oral body temperature | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of changes in vital signs as measured by heart rate, blood pressure, respiratory rate and oral body temperature reported
Changes in 12-lead ECG measures | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of changes in 12-ECG measures reported
Changes in physical examination measures | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of changes in physical examination measures reported
Changes in blood safety lab parameters | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of changes in blood safety parameters reported
Changes in urine safety lab parameters | Between Screening and 7 days after the last dosing
  To evaluate the safety and tolerability of GLPG1205 after multiple oral doses in healthy male subjects with or without coadministration of a cocktail of CYP450 substrates in terms of changes in urine safety parameters reported

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Desrivot J, Van Kaem T, Allamassey L, Helmer E. Effect of GLPG1205, a GPR84 Modulator, on CYP2C9, CYP2C19, and CYP1A2 Enzymes: In Vitro and Phase 1 Studies. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1007-1017. doi: 10.1002/cpdd.956. Epub 2021 May 6. PMID 33955686